CLINICAL TRIAL: NCT02492399
Title: Compare the Results for the Extended Myoectomy and Standard Morrow's Myoectomy in Patients With Ventricular Obstruction of the Left Ventricular Output
Brief Title: Comparisonof Extended Myoectomy and Myoectomy by Morrow in Patients With Hypertrophic Obstructive Cardiomyopathy (HOCM)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 12-435
Record Dates: First submitted 2015-07-01; First posted 2015-07-08 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Hypertrophic Obstructive Cardiomyopathy
Keywords: hypertrophic cardiomyopathy; mitral valve; SAM syndrome
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- myectomy by Morrow (Other): Procedure: myectomy by Morrow.
  Will be included in a group of 30 patients with obstructive hypertrophic cardiomyopathy and mitral insufficiency. In the case of conservation SAM syndrome and mediated mitral insufficiency, the result will be read as unsatisfactory. Patients will perform advanced myoectomy. All patients who need to be supplemented by the operation extension myoectomy subsequently run out in the second group. When it is impossible to eliminate mediated mitral regurgitation without mitral valve replacement, patients performed myoectomy and mitral valve replacement. The result in this case is read as completely unsatisfactory. Upon reaching 15% replacement mitral valve study terminated.
  Evaluation results will be made myoectomy as TEE and direct tensiometer.
  Interventions: Procedure: myectomy by Morrow
- extended myectomy (Other): Procedure: extended myectomy.
  Will be included in a group of 30 patients with obstructive hypertrophic cardiomyopathy and mitral insufficiency. Intraoperatively for all patients will be executed TEE to calculate the volume of excision. All patients will be performed extended myoectomy which supplemented resection and release of the papillary muscles. In case of unsatisfactory MV repair will reconnect the device artificial circulation and mitral valve replacement. The result in this case will become engrossed in reading as completely unsatisfactory. At achievement of 15% prosthetics of the mitralny valve research stops.
  Evaluation results will be made myoectomy as TEE and direct tensiometer .
  Interventions: Procedure: extended myectomy

INTERVENTIONS:
Procedure: extended myectomy — The scheme of extended septal myectomy: Two parallel incisions were made into the septal bulge and connected to remove the muscle mass. Myectomy was extended to the base of the papillary muscles, when midseptal thickening was present. The papillary muscles were grasped and pushed medially to visualize the abnormal connections between the papillary muscles and the anterior wall of the ventricle. A blade was used to divide the thickened abnormal attachments. A pituitary rongeur may be used to resect a portion of the junction of the papillary and lateral wall. This reduces the diameter of the papillary muscle and allows for posterior displacement of the anterior mitral leaflet. Division of abnormal attachments and thinning of the papillary muscles is critical for the treatment of SAM.
  Other Names: myectomy
  Arms: extended myectomy
Procedure: myectomy by Morrow — A first myotomy is made into the septum just below the base of the right coronary leaflet at a point 2-3 mm to the right of the commissure between the left and right coronary leaflets. A second myotomy is made in the same manner, parallel to the first one and about 1 cm to the right of it. The two vertical myotomies are made and cornnected transversely in the interventricular septum. The muscle bar is then grasped with the angled rongeur and the instrument is pushed firmly toward the apex, peeling the mtusele from its anterior septal attachments. After completion of the resectioni, a rectangular channel about 1 X 1.5 cm is palpable from the valve ring toward the apex for a dis- tance of about 4 cm.
  Other Names: myectomy
  Arms: myectomy by Morrow

SUMMARY:
The purpose of this study is to determine whether the application of the extended myoectomy in patients with obstruction of the left ventricular output more efficient than standard myoectomy by Morrow.

DETAILED DESCRIPTION:
Many years myoectomy for Morrow was the gold standard in the treatment of obstructive hypertrophic cardiomyopathy. Currently more retrospective data in the literature about the good results the extended septal myectomy. Use of extended myomectomy eliminates mitral insufficiency due to SAM syndrome. The question remains whether it is possible at hypertrophic cardiomyopathy basal part and mediated mitral insufficiency use only myoectomy by Morrow is achieved regression SAM syndrome and release output of the left ventricle. Planned to create two equal groups of 30 people that will use two methods of surgical treatment of obstructive hypertrophic cardiomyopathy. The study will be terminated in the event of complete AV block more than 2% and unsatisfactory results of a myoectomy requiring perform mitral valve replacement in more than 15% of the patients studied. The study assumed crossover: in case of failure elimination SAM syndrome and mediated mitral insufficiency myoectomy by Morrow for patients will perform extended myoectomy in the case of a good result in patients are moved to the second group.

Planned studies the long-term and immediate results of operations:

* Quantitative determination of enzymes of myocardial injury: creatine phosphokinase MB and troponin I.
* Determination of atrial natriuretic peptide (ANP) and brain natriuretic peptide (VNP).
* MRI with contrast heart to assess remodeling of the heart chambers and heart weight measurements.
* TEE evaluation function and mitral valve gradient at the output of the left ventricle.

ELIGIBILITY:
Inclusion Criteria:

* Able to sign Informed Consent and Release of Medical Information forms
* Age ≥ 18 years
* obstructive hypertrophic cardiomyopathy
* mediated mitral insufficiency by SAM syndrome
* II-IV (NYHA),
* average systolic pressure gradient greater than 50 mm Hg. Art. at rest;
* basal or medium ventricular obstruction

Exclusion Criteria:

* Related defect of the aortic valve;
* Organic mitral valve disease (dysplasia, rheumatic fever, infective endocarditis);
* Surgically significant coronary artery lesions;
* Patients requiring implantation of a cardioverter-defibrillator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The pressure gradient in the output section of the left ventricle | one year

SECONDARY OUTCOMES:
The function of the mitral valve | one year
  (Residual mitral regurgitation, SAM syndrome)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandr V Bogachev-Prokophiev, PhD, Principal Investigator — Meshalkin Research Institute of Pathology of Circulation
Locations (1):
- Novosibirsk State Research Institute of Circulation Pathology, Novosibirsk, Novosibirsk Territory, Russia